CLINICAL TRIAL: NCT06361810
Title: A Phase 1/2 Open-label Study of Pembrolizumab Combined With PNT-2002 Radioligand Therapy in Patients With Metastatic Renal Cell Carcinoma
Brief Title: PSMA Therapy and Immunotherapy in Kidney Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: funding withdrawn
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00430008
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Renal Cell Carcinoma; Metastatic Clear Cell Renal Cell Carcinoma
Keywords: Kidney Cancer; Pembrolizumab; 177Lu-PNT2002; Pylarify
MeSH Terms: conditions — Carcinoma, Renal Cell; Clear-cell metastatic renal cell carcinoma; Kidney Neoplasms | interventions — pembrolizumab; 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 177Lu-PNT2002 3.4 GBq (Experimental): 177Lu-PNT2002 administered at 3.4 GBq intravenously (IV) every 8 weeks combined with the standard dose of pembrolizumab 400 mg IV every 6 weeks. 18F-DCFPyL administered as a single bolus intravenous radioactive dose injection of 333 megabecquerel (MBq) (9 mCi) at screening, week 12 and week 24.
  Interventions: Drug: Pembrolizumab; Drug: 177Lu-PNT2002; Drug: (F-18)-DCFPyL
- 177Lu-PNT2002 5.1 GBq (Experimental): 177Lu-PNT2002 administered at 5.1 GBq intravenously (IV) every 8 weeks combined with the standard dose of pembrolizumab 400 mg IV every 6 weeks. 18F-DCFPyL administered as a single bolus intravenous radioactive dose injection of 333 MBq (9 mCi) at screening, week 12 and week 24.
  Interventions: Drug: Pembrolizumab; Drug: 177Lu-PNT2002; Drug: (F-18)-DCFPyL
- 177Lu-PNT2002 6.8 GBq (Experimental): 177Lu-PNT2002 administered at 6.8 GBq intravenously (IV) every 8 weeks combined with the standard dose of pembrolizumab 400 mg IV every 6 weeks. 18F-DCFPyL administered as a single bolus intravenous radioactive dose injection of 333 MBq (9 mCi) at screening, week 12 and week 24.
  Interventions: Drug: Pembrolizumab; Drug: 177Lu-PNT2002; Drug: (F-18)-DCFPyL
- Dose Expansion (Experimental): 177Lu-PNT2002 administered at the maximum tolerated dose (determined by the 3 dose levels in the dose escalation phase of the study) intravenously (IV) every 8 weeks combined with the standard dose of pembrolizumab 400 mg IV every 6 weeks. 18F-DCFPyL administered as a single bolus intravenous radioactive dose injection of 333 MBq (9 mCi) at screening, week 12 and week 24.
  Interventions: Drug: Pembrolizumab; Drug: 177Lu-PNT2002; Drug: (F-18)-DCFPyL

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be administer at 400 mg IV every 6 weeks in combination with 177Lu-PNT2002 until the maximum tolerated dose of 177Lu-PNT2002 is reached during the dose escalation phase.
  Pembrolizumab will be administer at 400 mg IV every 6 weeks for a maximum of 17 cycles (6 weeks in each cycle) during the dose expansion phase.
  Other Names: Keytruda
Drug: 177Lu-PNT2002 — 177Lu-PNT2002 given intravenously every 8 weeks will be administered at 3.4 GBq, 6.1 Gbq, or 6.8 Gbq in combination with the standard dose of pembrolizumab 400 mg given intravenously every 6 weeks until the maximum tolerated dose is reached during the dose escalation phase.
  177Lu-PNT2002 given intravenously every 8 weeks will be administered at the determined maximum tolerated dose for a maximum of 4 cycles in combination with the standard dose of pembrolizumab 400 mg given intravenously every 6 weeks for a maximum of 17 cycles.
  Other Names: 177Lu-PSMA I&T
Drug: (F-18)-DCFPyL — Patients will be administered 18F-DCFPyL as a single bolus intravenous radioactive dose injection of 333 MBq (9 mCi) at screening, week 12 and week 24.
  Other Names: Pylarify

SUMMARY:
This is a multi-center, single arm open label phase 1b/2 study of pembrolizumab in combination with 177Lu-PNT2002 (also known as 177Lu-PSMA I&T) radiopharmaceutical therapy in patients with metastatic clear cell renal cell carcinoma (RCC) who have progressed after prior treatment with anti-programmed cell death protein 1 (PD1) or PD-L1 immune-checkpoint inhibitors (ICIs). The study comprises 2 phases: an open-label Phase 1b dose escalation portion followed by a Phase 2 dose expansion portion. Investigators hypothesize that pembrolizumab in combination with 177Lu-PNT2002 in in patients with metastatic clear cell RCC at a biologically active dose will result in tolerable safety profile and it will lead to improved radiological objective responses in patients who have progressed after prior treatment with standard anti-PD1 or anti- Programmed Cell Death Ligand 1 (PDL1) immune-checkpoint inhibitor containing regimen when compared to historic controls. Patients in both phases will have prostate-specific membrane antigen (PSMA), positron emission tomography (PET) imaging with the radiotracer (F-18)-DCFPyl, to help detect any spread of the cancer.

DETAILED DESCRIPTION:
In the dose escalation phase, three dose levels of 177Lu-PNT2002 given intravenously every 8 weeks, starting from 3.4 gigabequerel (GBq) in combination with the standard dose of pembrolizumab 400 mg given intravenously every 6 weeks. After determining the maximum tolerated dose (MTD) or the recommended Phase 2 Dose (RP2D), the study will proceed to the dose expansion phase and in this portion of the study, patients will receive 177Lu-PNT-2002 intravenously every 8 weeks at the MTD/RP2D for a maximum of 4 cycles in combination pembrolizumab 400 mg intravenously every 6 weeks for a maximum of 17 cycles.

The primary objective of the phase 1b portion of the study is to determine the MTD or RP2D of 177Lu-PNT2002 radiopharmaceutical therapy in combination with pembrolizumab in patients with metastatic clear cell RCC. The primary objective of the phase 2 portion of the study is to evaluate the efficacy of 177Lu-PNT2002 in combination with pembrolizumab in patients with metastatic clear cell RCC who progressed on prior anti PD-1/PDL1 therapy based on objective response rate (ORR) by RECIST 1.1 criteria.

Patients in both phases will receive PSMA-PET with (F-18)-DCFPyl at screening, 12 weeks, and 24 weeks. (F-18)-DCFPyl was developed as a diagnostic radiotracer for the detection of prostate cancer and was FDA approved in 2021 for the detection of PSMA positive lesions in men with prostate cancer. However, PSMA is not entirely prostate-specific, as it has been shown to be present on neovascular endothelium of numerous solid tumors, including RCC. Prior studies have demonstrated high sensitivity and specificity of the detection of metastatic clear cell RCC lesions using PET imaging with various PSMA radiotracers, such as (F-18)-DCFPyl. Based on this, the high expression of PSMA in RCC and the synergy of PSMA radiopharmaceuticals with ICIs, such as pembrolizumab, provide a novel treatment strategy in RCC.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of clear cell RCC will be enrolled in this study.
2. Participants must have progressed on treatment with an anti-PD-1/L1 ICI administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria:

   1. Treatment with at least 6 weeks of an approved anti-PD-1/L1 ICI.
   2. More than one prior line of anti-PD-1/L1 ICI is allowed.
   3. The immediate prior line of therapy is not mandated to be with anti-PD-1/L1 ICI.
   4. Postoperative or adjuvant systemic therapy can be counted as a prior ICI therapy as long as recurrence is detected within 6 months of completion of treatment, in which case it will be counted as a prior therapy for metastatic disease.
3. Metastatic or locally advanced inoperable clear cell RCC.
4. Participants who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline.
5. Evidence of positive PSMA avid lesions as per (F-18)-DCFPyL PSMA PET scan at screening. Positive lesions on PSMA-PET are defined as those with maximum standardized uptake value (SUVmax) values greater than liver as assessed by the local site investigator radiologist.
6. At least 70% of all the following lesions must PSMA-PET positive:

   1. Lymph nodes that measure ≥ 25 mm in short axis on anatomic imaging.
   2. Bone metastasis with soft tissue component ≥ 10 mm in short axis.
   3. Solid organ metastasis ≥ 10 mm in short axis.
7. A maximum of 4 prior lines of systemic therapy is allowed, including more than one line of ICI regimens.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 with a life expectancy ≥ 6 months
9. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
10. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
11. Female subjects of childbearing potential must be non-pregnant, non-lactating, and have a urine or serum pregnancy test within 24 hours prior to administration of each PNT-2002 dose.
12. Females of childbearing potential who are sexually active with a non-sterilized male partner agree to use effective methods of contraception from screening, throughout the study treatment and agree to continue using such precautions for 4 months after the final dose of study drug.
13. Non-sterilized males who are sexually active with a female of childbearing potential must agree to use effective methods of contraception from Day 1 throughout the study treatment and for 6 months after the final dose of study drug.
14. Have adequate organ function. Blood Specimens must be collected within 7 days prior to the start of study intervention.

Exclusion Criteria:

1. Renal cell carcinoma with non-clear cell histology.
2. Prior exposure to radioligand therapy or radioisotope therapy.
3. Treatment with RCC standard of care anti-cancer therapy within 14 days prior to initiation of study treatment
4. Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
5. PSMA targeted imaging within 2 weeks prior to screening.
6. Has received prior radiotherapy within 2 weeks of start of study intervention or radiation-related toxicities requiring corticosteroids. Note: Two weeks or fewer of palliative radiotherapy for non-central nervous system diseases permitted. The last radiotherapy treatment must have been performed at least 7 days before the first dose of study intervention.
7. Must have recovered from any grade 3 or higher reversible toxicity to prior anti cancer therapy treatments.
8. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
9. Has a diagnosis of immunodeficiency (e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV) or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
10. Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded. Participants with low-risk early-stage prostate cancer (T1-T2a, Gleason score ≤6, and prostate-specific antigen (PSA) <10 ng/mL) either treated with definitive intent or untreated in active surveillance with stable disease are not excluded.
11. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
12. Has severe hypersensitivity (≥Grade 3) to pembrolizumab or (F-18)-DCFPyL (Pylarify) and/or any of their components.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid)
14. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
15. Has an active infection requiring systemic therapy
16. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable (HBV) DNA and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.

    Note: Hepatitis B and C screening tests are not required unless:

    Known history of hepatitis B virus (HBV) and hepatitis C virus (HCV) infection As mandated by local health authority
17. Has not adequately recovered from major surgery or has ongoing surgical complications.
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
20. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
21. Has had an allogenic tissue/solid organ transplant.
22. Known history of HIV infection. HIV testing is not required unless mandated by local health authority.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Safety assessed by the incidence of dose limiting toxicities. | Day 28
  Number of incidences of dose limiting toxicities during days 1 to 28 of cycle 1.
Objective response rate by RECIST 1.1 criteria | 3 years post therapy initiation
  Proportion of patients with an objective response, defined as Complete Response or Partial Response by RECIST 1.1. Dose expansion phase of the trial.

SECONDARY OUTCOMES:
Progression free survival | 4 years post therapy initiation
  Median time to progression free survival of participants on study therapy. Dose escalation phase of the trial.
Safety as assessed by number of participants experiencing adverse events | 2 years post therapy initiation
  Number of participants who experience adverse events Grade 3-5, as defined by Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Dose escalation phase of the trial.
Disease control rates | 3 years post therapy initiation
  Proportion of participants with Partial Response, Complete Response, or Stable Disease for six months or more. Dose expansion phase of the trial.
Duration of response to study therapy | 3 years post therapy initiation
  Time from the start of a Complete Response or Partial Response to progression or death. Dose expansion phase of the trial.
Overall survival rate | 4 years post therapy initiation
  Proportion of participants who complete the survival follow-up visits. Dose expansion phase of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Ged, MD, Principal Investigator — Johns Hopkins University